CLINICAL TRIAL: NCT04019223
Title: The Diagnostic Performance of Anti-Tissue Transglutaminase IgA Antibodies Serum Level for Detection of Patients With Celiac Disease
Brief Title: Anti-Tissue Transglutaminase IgA Antibodies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Suzan Alaa Babran, principal Investigator, Assiut University
Other Study IDs: DPAAB
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Celiac Disease in Children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anti-tissue transglutaminase group: serum IgA-tissue transglutaminase antibody (tTG) was analyzed in serum using a quantitative automated ELISA method by means of a commercially available detection kit using recombinant human tTG as antigen recommended cut-off by the manufacturer > 8 U/mL).
  Interventions: Diagnostic Test: anti-tissue transglutaminase group; Diagnostic Test: biopsy group
- biopsy group: upper gastrointestinal endoscopic examination will be done and the jejunal histopathological examinations will be done at the Histopathology Laboratory. The features consistent with CD included: hyperplasia of crypts, atrophy of villous, and increase of intraepithelial lymphocytes.Duodenal samples will be processed using haematoxylin/eosin staining and CD3 immunophenotyping. The number of intra-epithelial lymphocytes (IEL), the architecture of villi, and the inflammatory cell infiltration of the lamina propria will be assessed. Histopathological changes will be classified according to the Marsh-Oberhuber criteria.Lymphocytic enteropathy (Marsh 1 lesion) was defined as 25 or more IEL per 100 epithelial nuclei, and normal villous architecture.
  Interventions: Diagnostic Test: anti-tissue transglutaminase group; Diagnostic Test: biopsy group

INTERVENTIONS:
Diagnostic Test: anti-tissue transglutaminase group — Determination of anti-tissue transglutaminase IgA antibodies serum level.
Diagnostic Test: biopsy group — Intestinal biopsy for histopathology study the jejunal histopathological

SUMMARY:
Celiac disease is the most common genetically related food intolerance, worldwide. It is an immune mediated intolerance to gluten (from wheat, barley, or rye) in genetically susceptible individuals .The disease primarily affects the small intestine, where it progressively leads to flattening of the small intestinal mucosa .

DETAILED DESCRIPTION:
Within this definition, patients can further be defined as having silent, potential, or latent celiac disease. The term silent celiac disease refers to patients fulfilling the definition above, but presenting no symptoms. Typically, such diagnoses are made by screening asymptomatic individuals, who are at increased risk for celiac disease. The term potential celiac disease describes patients who have specific serum autoantibodies and may or may not have symptoms consistent with celiac disease, but lack evidence of the autoimmune damage to the intestinal mucosa. A final category of celiac patients is represented by the so-called latent celiac disease: individuals with normal mucosal morphology (like the potential) but known to have had a gluten-dependent enteropathy at some point in their life .

Malabsorption results from injury to the small intestine with loss of absorptive surface area, reduction of digestive enzymes, and consequential impaired absorption of micronutrients such as fat-soluble vitamins, iron and potentially B12 and folic acid. In addition, the inflammation exacerbates symptoms of malabsorption by causing net secretion of fluid that can result in diarrhea. The failure of absorption of adequate calories leads to weight loss, and the malabsorption results in abdominal pain and bloating .

A positive family history is a risk factor for celiac disease. The frequency of celiac disease is higher among first- and second-degree relatives of persons with celiac disease, although prevalence estimates range from 5 to 20 percent . Frequency of celiac disease is also higher among persons with other autoimmune diseases, such as type 1 diabetes mellitus, inflammatory luminal gastrointestinal disorders, Down syndrome, Turner's syndrome, IgA deficiency, and IgA nephropathy .

Gastrointestinal and extra-intestinal manifestations of celiac disease include diarrhea, abdominal pain, abdominal distention, anorexia, vomiting, constipation, failure to thrive, chronic fatigue, anemia, osteoporosis, aphthous stomatitis, elevated liver enzymes, joint/muscle pain, epilepsy, and peripheral neuropathy .

Clinical practice guidelines recommend to starting with the serum anti-tissue transglutaminase IgA antibodies (anti-tTG IgA) test as a diagnostic testing for celiac disease. The tTG IgA test is the standard method of testing for celiac disease . Clinical practice in guidelines the United States and Europe recommend intestinal biopsy to confirm the diagnosis of celiac disease (e.g., based on presence of villous atrophy hyperplasia of crypts, and increase of intraepithelial lymphocytes) and to distinguish celiac disease from other disorders affecting the small intestine. Intestinal biopsy may also be performed if clinical suspicion for celiac disease is high but serologic tests are negative . It has been suggested that a combination of serologic tests could be used to establish celiac disease diagnosis as an alternative to biopsy, but it is unclear how frequently celiac disease is diagnosed in the absence of biopsy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* • patients with symptoms suggestive of celiac disease

Exclusion Criteria:

•chronic active gastrointestinal disease, i.e., irritable bowel syndrome inflammatory bowel disease .

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients in this research will be subjected to :
  Besides meticulous history and thorough clinical examination, all the cases will be subjected to the following investigations :
  * Complete blood count.
  * Determination of electrolytes serum levels: Na, K, Mg, Ca and Ph.
  * Liver function tests.
  * Determination of anti-tissue transglutaminase IgA antibodies serum level.
  * Intestinal biopsy for histopathology study the jejunal histopathological
  * examinations will be done at the Histopathology Laboratory.
  * The features consistent with CD included: hyperplasia
  * of crypts, atrophy of villous, and increase of intraepithelial
  * lymphocytes.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
measure of Anti- tissue will be performed to calculate the post-test probability of celiac disease. | within 24 hours
  tTG are regarded as qualitative, i.e., positive or negative.Values of tTG between 2 and 7 U/mL will be considered as doubtful positive, and those of 7 U/mL or more as positive.
  cut-off of ≥7 U/mL will be used in this study.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richey R, Howdle P, Shaw E, Stokes T; Guideline Development Group. Recognition and assessment of coeliac disease in children and adults: summary of NICE guidance. BMJ. 2009 May 27;338:b1684. doi: 10.1136/bmj.b1684. No abstract available. PMID 19474030
- [Result] Sansotta N, Amirikian K, Guandalini S, Jericho H. Celiac Disease Symptom Resolution: Effectiveness of the Gluten-free Diet. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):48-52. doi: 10.1097/MPG.0000000000001634. PMID 28514243
- [Result] Burgin-Wolff A, Mauro B, Faruk H. Intestinal biopsy is not always required to diagnose celiac disease: a retrospective analysis of combined antibody tests. BMC Gastroenterol. 2013 Jan 23;13:19. doi: 10.1186/1471-230X-13-19. PMID 23343249
- [Result] Fasano A, Berti I, Gerarduzzi T, Not T, Colletti RB, Drago S, Elitsur Y, Green PH, Guandalini S, Hill ID, Pietzak M, Ventura A, Thorpe M, Kryszak D, Fornaroli F, Wasserman SS, Murray JA, Horvath K. Prevalence of celiac disease in at-risk and not-at-risk groups in the United States: a large multicenter study. Arch Intern Med. 2003 Feb 10;163(3):286-92. doi: 10.1001/archinte.163.3.286. PMID 12578508
- [Result] Godfrey JD, Brantner TL, Brinjikji W, Christensen KN, Brogan DL, Van Dyke CT, Lahr BD, Larson JJ, Rubio-Tapia A, Melton LJ 3rd, Zinsmeister AR, Kyle RA, Murray JA. Morbidity and mortality among older individuals with undiagnosed celiac disease. Gastroenterology. 2010 Sep;139(3):763-9. doi: 10.1053/j.gastro.2010.05.041. Epub 2010 Jun 1. PMID 20685275
- [Result] Murray JA. Celiac disease in patients with an affected member, type 1 diabetes, iron-deficiency, or osteoporosis? Gastroenterology. 2005 Apr;128(4 Suppl 1):S52-6. doi: 10.1053/j.gastro.2005.02.029. PMID 15825127
- [Result] Rubio-Tapia A, Hill ID, Kelly CP, Calderwood AH, Murray JA; American College of Gastroenterology. ACG clinical guidelines: diagnosis and management of celiac disease. Am J Gastroenterol. 2013 May;108(5):656-76; quiz 677. doi: 10.1038/ajg.2013.79. Epub 2013 Apr 23. PMID 23609613
- [Result] Rubio-Tapia A, Ludvigsson JF, Brantner TL, Murray JA, Everhart JE. The prevalence of celiac disease in the United States. Am J Gastroenterol. 2012 Oct;107(10):1538-44; quiz 1537, 1545. doi: 10.1038/ajg.2012.219. Epub 2012 Jul 31. PMID 22850429